CLINICAL TRIAL: NCT06490900
Title: Influence of One Session of Intermittent Hypoxia on Glycemic Control
Brief Title: Influence of Intermittent Hypoxia on Glycemic Control
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas at Austin (Other)
Responsible Party: Principal Investigator, Sophie Lalande, Assistant Professor, University of Texas at Austin
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 2020050108
Record Dates: First submitted 2024-06-29; First posted 2024-07-08 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2025-03

CONDITIONS: Hypoxemia
MeSH Terms: conditions — Hypoxia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intermittent hypoxia (Experimental): The intermittent hypoxia protocol will consist of eight 4-minute hypoxic cycles (arterial oxygen saturation of 80%) interspersed with normoxic cycles (room air) to resaturation.
  Interventions: Behavioral: Intermittent hypoxia
- Intermittent normoxia (Sham Comparator): The intermittent normoxia protocol will consist of eight 4-minute normoxic cycles (compressed air) interspersed with 1-minute normoxic cycles (room air).
  Interventions: Behavioral: Intermittent normoxia

INTERVENTIONS:
Behavioral: Intermittent hypoxia — The intermittent hypoxia protocol will consist of eight 4-minute hypoxic cycles (arterial oxygen saturation of 80%) interspersed with normoxic cycles (room air) to resaturation.
  Arms: Intermittent hypoxia
Behavioral: Intermittent normoxia — The intermittent normoxia protocol will consist of eight 4-minute normoxic cycles (compressed air) interspersed with 1-minute normoxic cycles (room air).
  Arms: Intermittent normoxia

SUMMARY:
The aim of this research project is to determine the effect of intermittent hypoxia on glucose uptake in response to an oral glucose tolerance test in healthy individuals, individuals with prediabetes and patients with type 2 diabetes.

DETAILED DESCRIPTION:
For the past 100 years, cardiovascular disease has been the leading cause of death in the United States. An aging population, increasing levels of obesity and the predominance of a sedentary lifestyle contribute to the growing incidence of type 2 diabetes, one of the major modifiable risk factors for cardiovascular disease. It is now predicted that 1 in 3 adults will develop diabetes by 2050, implying that a large percentage of the population will become at high risk for cardiovascular disease, the most common cause of death in patients with type 2 diabetes. While exercise reduces insulin resistance and the elevated glucose levels associated with type 2 diabetes, only 28% of the adult population with diabetes meet physical activity recommendations. Thus, our overall objective is to identify an alternative, non-pharmacological intervention that prevents the development of type 2 diabetes in individuals with prediabetes, and treats the insulin resistance and hyperglycemia in patients already diagnosed with type 2 diabetes.

The Nobel Prize in Physiology was recently awarded to scientists who established the basis for our understanding of how varying oxygen levels affect cellular metabolism, which paved the way for promising new strategies to fight diseases. Breathing low levels of oxygen, or hypoxia, stimulates glucose uptake in skeletal muscle via 5' adenosine monophosphate-activated protein kinase (AMPK), the same signaling pathway as muscle contraction, which acts independently from the actions of insulin. Thus, patients with type 2 diabetes were exposed to either normoxia or 60 min of continuous hypoxia (fraction of inspired oxygen of ~0.15, arterial oxygen saturation of 92%) immediately before performing a 4-hour intravenous glucose tolerance test. Hypoxia lowered blood glucose levels and did not affect insulin concentrations, therefore, it was suggested that the improved glycemic control was caused by the activation of the AMPK pathway in combination with an improved insulin sensitivity. Similarly, a single exposure to intermittent hypoxia, consisting of 6 min at a fraction of inspired oxygen of 0.13 alternated with 6 min of normoxia for 1 hour, improved glycemic control in patients with type 2 diabetes. Specifically, there was a greater decrease in glucose levels measured immediately after intermittent hypoxia, and the increase in glucose levels following a meal was attenuated following intermittent hypoxia when compared to a placebo condition. A decrease in glucose levels was also observed following a single session of intermittent hypoxia, consisting of brief desaturation and resaturation cycles to maintain an arterial oxygen saturation of 80% for approximately 70 min, in overweight and obese individuals with normal baseline glucose levels.

The specific aim of this research project is to identify whether exposure to intermittent hypoxia during an oral glucose tolerance test attenuates the increase in glucose levels in healthy individuals, individuals with prediabetes and patients with type 2 diabetes. It is hypothesized that exposure to intermittent hypoxia will attenuate the increase in glucose levels in response to an oral glucose tolerance test in healthy individuals, individuals with prediabetes and patients with type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged 18 to 80 years old

Exclusion Criteria:

* Have uncontrolled stage 2 hypertension (˃140/90 mmHg)
* Are smokers
* Are pregnant
* Have a history of cardiovascular disease or indication of cardiovascular disease such as myocardial infarction, left ventricular hypertrophy, ischemic heart disease (or prior ischemia), stroke, and/or other vascular disease
* Have a history of lung disease
* Are taking insulin or more than one antihypertensive medication
* Have poorly controlled diabetes: HbA1c levels ˃ 9%
* Have been previously diagnosed with diabetic complications (nephropathy, neuropathy, retinopathy) by their family doctor

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2021-02-05 (Actual); Primary Completion 2024-03-03 (Actual); Study Completion 2024-11-26 (Actual)

PRIMARY OUTCOMES:
Change in plasma glucose levels | Collected at minutes 0, 30, 60, 90 and 120 of the oral glucose tolerance test
  Plasma glucose levels obtained from a venous catheter during a 2-hour oral glucose tolerance test

CONTACTS AND LOCATIONS:
Overall Officials: Sophie Lalande, Principal Investigator — UT Austin
Locations (1):
- The Unviersity of Texas at Austin, Austin, Texas, United States